CLINICAL TRIAL: NCT04950127
Title: A Two-part, Randomized, Placebo Controlled, Double Blind, Multicenter, Phase 3 Study to Evaluate the Efficacy and Safety of Linerixibat for the Treatment of Cholestatic Pruritus in Participants With Primary Biliary Cholangitis (PBC)
Brief Title: Global Linerixibat Itch Study of Efficacy and Safety in Primary Biliary Cholangitis (PBC) (GLISTEN)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 212620
Expanded Access: NCT05448170 (Available)
Record Dates: First submitted 2021-06-25; First posted 2021-07-06 (Actual); Results first posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Pruritus
Keywords: Cholestasis; GLISTEN; GSK2330672; Itch; Primary biliary cholangitis; Pruritus
MeSH Terms: conditions — Pruritus; Cholestasis; Liver Cirrhosis, Biliary

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive linerixibat and/or placebo during the study.
Who Masked: Participant, Investigator
Masking Description: Participants and investigator will be blinded to the study treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part A: Linerixibat 40 milligrams (mg) (Experimental): Participants were randomized to receive linerixibat 40 mg tablet orally twice a day (BID) in Part A (up to Week 24).
  Interventions: Drug: Linerixibat
- Part A: Placebo (Experimental): Participants were randomized to receive Placebo orally twice a day (BID) in Part A (up to Week 24).
  Interventions: Drug: Linerixibat; Drug: Placebo
- Part B: Placebo in Part A and Part B (Placebo Comparator): Participants who were randomized to receive Placebo (up to Week 24) orally twice a day (BID) in Part A, continued to receive Placebo (from Week 24 to Week 32) orally twice a day (BID) in Part B.
  Interventions: Drug: Placebo
- Part B: Placebo in Part A and Linerixibat 40 mg in Part B (Experimental): Participants who were randomized to receive Placebo (up to Week 24) orally twice a day (BID) in Part A, switched to receive linerixibat 40 mg tablet orally twice a day (BID) (from Week 24 to Week 32) in Part B.
  Interventions: Drug: Linerixibat; Drug: Placebo
- Part B: Linerixibat 40 mg in Part A and Placebo in Part B (Experimental): Participants who were randomized to receive linerixibat 40 mg tablet orally BID (up to Week 24) in Part A, switched to receive Placebo (from Week 24 to Week 32) orally twice a day (BID) in Part B.
  Interventions: Drug: Linerixibat; Drug: Placebo
- Part B: Linerixibat 40 mg in Part A and Part B (Experimental): Participants who were randomized to receive linerixibat 40 mg tablet orally twice a day (BID) (up to Week 24) in Part A, continued to receive linerixibat 40 mg twice a day (BID) (from Week 24 to Week 32) in Part B.
  Interventions: Drug: Linerixibat

INTERVENTIONS:
Drug: Linerixibat — Participants will receive linerixibat.
  Arms: Part A: Linerixibat 40 milligrams (mg); Part A: Placebo; Part B: Linerixibat 40 mg in Part A and Part B; Part B: Linerixibat 40 mg in Part A and Placebo in Part B; Part B: Placebo in Part A and Linerixibat 40 mg in Part B
Drug: Placebo — Participants will receive placebo.
  Arms: Part A: Placebo; Part B: Linerixibat 40 mg in Part A and Placebo in Part B; Part B: Placebo in Part A and Linerixibat 40 mg in Part B; Part B: Placebo in Part A and Part B

SUMMARY:
This is a 2-part study in PBC participants with cholestatic pruritus and will evaluate the efficacy, safety and impact on health-related quality of life of linerixibat compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants must be between 18 to 80 years of age inclusive, at the time of signing the informed consent.
* Participants who have documented PBC.
* Participants who have moderate to severe itch.

Exclusion Criteria:

* Total bilirubin >2.0 times Upper Limit of Normal (ULN) using the average of two Baseline measures.
* Screening Alanine Aminotransferase (ALT) > 6 times ULN in a single Baseline measure or ALT > 5 times ULN using the average of two Baseline measures.
* Screening estimated glomerular filtration rate (eGFR) <30 milliliter per minute per 1.73 square meter (mL/min/1.73m^2).
* History or presence of hepatic decompensation (e.g., variceal bleeding, hepatic encephalopathy or ascites).
* Presence of HBsAg positive hepatitis B or hepatitis C (HCV) (anti-HCV and Ribonucleic acid [RNA] detected) infection, primary sclerosing cholangitis (PSC), alcoholic liver disease and/or confirmed hepatocellular carcinoma or biliary cancer.
* Current clinically significant diarrhea or active inflammatory ileal disease according to Investigator´s clinical judgment.
* Current symptomatic cholelithiasis or cholecystitis.
* Current diagnosis of primary skin disorders with itch as a characteristic feature (e.g., atopic dermatitis, psoriasis).
* Primary sleep disorders such as but are not limited to sleep apnea, narcolepsy, hypersomnia.
* Initiation, discontinuation or change in dose of ursodeoxycholic acid (UDCA), bezafibrate or fenofibrate in the 8 weeks prior to Screening.
* Use of obeticholic acid: within 8 weeks prior to Screening. (Participants may not initiate or restart during the study).
* Initiation, discontinuation, or change in dose of any of the following in the 8 weeks prior to Screening: bile acid binding resins, rifampicin, naltrexone, naloxone, nalfurafine, pregabalin, gabapentin, sertraline or other selective serotonin reuptake inhibitor (SSRIs), antihistamines used for the treatment of itching.
* Administration of any other human ileal bile acid transporter (IBAT) inhibitor in the 12 weeks prior to screening.
* Any planned procedures intended to treat cholestatic pruritus such as nasobiliary drainage or ultraviolet light therapy from Screening and throughout the study.
* History of sensitivity or intolerance to the study treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2024-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (103):
- United States (16):
  - GSK Investigational Site, Davis, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Hialeah, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Jackson, Mississippi
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Morrisville, North Carolina
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
- Argentina (7):
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Capital Federal
  - GSK Investigational Site, Ciudad AutOnoma de Buenos Aire
  - GSK Investigational Site, Ciudad Autonoma de Bueno
  - GSK Investigational Site, Rosario
  - GSK Investigational Site, San Nicolás
  - GSK Investigational Site, Santa Fe
- GSK Investigational Site, Ghent, Belgium
- Brazil (4):
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
  - GSK Investigational Site, Botucatu
  - GSK Investigational Site, Brasília
  - GSK Investigational Site, Salvador
- Bulgaria (2):
  - GSK Investigational Site, Plovdiv
  - GSK Investigational Site, Sofia
- Canada (2):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Toronto, Ontario
- China (9):
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Changchun
  - GSK Investigational Site, Chongqing
  - GSK Investigational Site, Guangzhou
  - GSK Investigational Site, Nanchang
  - GSK Investigational Site, Nanjing
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Tianjin
  - GSK Investigational Site, Zhanjiang
- Czechia (3):
  - GSK Investigational Site, Ostrava
  - GSK Investigational Site, Pilsen
  - GSK Investigational Site, Prague
- France (4):
  - GSK Investigational Site, Créteil
  - GSK Investigational Site, Grenoble
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Paris
- Germany (3):
  - GSK Investigational Site, Erlangen
  - GSK Investigational Site, Essen
  - GSK Investigational Site, Münster
- GSK Investigational Site, Athens, Greece
- Israel (6):
  - GSK Investigational Site, Beersheba
  - GSK Investigational Site, Haifa
  - GSK Investigational Site, Holon
  - GSK Investigational Site, Jerusalem
  - GSK Investigational Site, Nahariya
  - GSK Investigational Site, Rehovot
- Italy (8):
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Modena
  - GSK Investigational Site, Monza
  - GSK Investigational Site, Napoli
  - GSK Investigational Site, Negrar Verona
  - GSK Investigational Site, Palermo
  - GSK Investigational Site, Roma
  - GSK Investigational Site, Rozzano MI
- Japan (12):
  - GSK Investigational Site, Ehime
  - GSK Investigational Site, Fukui
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Kagawa
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Nagano
  - GSK Investigational Site, Nagasaki
  - GSK Investigational Site, Nara
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokyo
- Mexico (2):
  - GSK Investigational Site, Mexico City
  - GSK Investigational Site, Monterrey
- Poland (5):
  - GSK Investigational Site, Częstochowa
  - GSK Investigational Site, Katowice
  - GSK Investigational Site, Mysłowice
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wroclaw
- Russia (4):
  - GSK Investigational Site, Kemerovo
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Novosibirsk
  - GSK Investigational Site, Samara
- Spain (3):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Seville
- United Kingdom (11):
  - GSK Investigational Site, Basingstoke
  - GSK Investigational Site, Cambridge
  - GSK Investigational Site, Durham
  - GSK Investigational Site, Hull
  - GSK Investigational Site, Liverpool
  - GSK Investigational Site, London
  - GSK Investigational Site, Newcastle upon Tyne
  - GSK Investigational Site, Plymouth
  - GSK Investigational Site, Reading Berkshire
  - GSK Investigational Site, Southampton
  - GSK Investigational Site, Surrey

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Hirschfield GM, Bowlus CL, Jones DEJ, Kremer AE, Mayo MJ, Tanaka A, Andreone P, Jia J, Jin Q, Macias-Rodriguez RU, Cobitz AR, Currie BM, Gorey C, Lazic I, Podmore D, Ribeiro A, Shannon JB, Swift B, McLaughlin MM, Levy C; GLISTEN Study Group. Linerixibat in patients with primary biliary cholangitis and cholestatic pruritus (GLISTEN): a randomised, multicentre, double-blind, placebo-controlled, phase 3 trial. Lancet Gastroenterol Hepatol. 2026 Jan;11(1):22-33. doi: 10.1016/S2468-1253(25)00192-X. Epub 2025 Oct 28. PMID 41173016
- [Derived] Carreno F, Karatza E, Mehta R, Collins J, Austin D, Swift B. Population Dose-Response-Time Analysis of Itch Reduction and Patient-Reported Tolerability Supports Phase III Dose Selection for Linerixibat. Clin Pharmacol Ther. 2024 Feb;115(2):288-298. doi: 10.1002/cpt.3103. Epub 2023 Dec 3. PMID 37953500

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 238 participants from Europe, North America, Latin America and Asia were enrolled and randomized.
Pre-assignment Details: This study was conducted in 2 parts: Part A and Part B. Participants were randomized in 1:1:1:1 ratio to receive either: linerixibat 40 milligram (mg) twice a day (BID) in Part A and Part B, linerixibat 40mg twice a day (BID) in Part A and placebo in Part B, placebo in Part A and Part B, or placebo in Part A and linerixibat 40mg twice a day (BID) in Part B.
Period: Part A (Day 1 to Week 24)
Arm/Group | Part A: Linerixibat 40 Milligrams (mg) | Part A: Placebo | Part B: Placebo in Part A and Part B | Part B: Placebo in Part A and Linerixibat 40 mg in Part B | Part B: Linerixibat 40 mg in Part A and Placebo in Part B | Part B: Linerixibat 40 mg in Part A and Part B
Started (Intent-to-Treat (ITT) Population: All participants randomly assigned to study treatment.) | 119 | 119 | 0 | 0 | 0 | 0
Safety Population (Safety Population: All randomized participants who take at least 1 dose of study intervention. Participants will be analyzed according to the treatment they actually received.) | 119 | 118 | 0 | 0 | 0 | 0
Completed | 103 | 108 | 0 | 0 | 0 | 0
Not Completed | 16 | 11 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 4 | 2 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 3 | 2 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 9 | 7 | 0 | 0 | 0 | 0
Period: Part B (Week 24 to Week 32)
Arm/Group | Part A: Linerixibat 40 Milligrams (mg) | Part A: Placebo | Part B: Placebo in Part A and Part B | Part B: Placebo in Part A and Linerixibat 40 mg in Part B | Part B: Linerixibat 40 mg in Part A and Placebo in Part B | Part B: Linerixibat 40 mg in Part A and Part B
Started (ITT Population of Part B included all participants who completed the Part A.) | 0 | 0 | 55 (Participants continued from Part A.) | 53 (Participants continued from Part A) | 49 (Participants continued from Part A) | 54 (Participants continued from Part A)
Safety Population (Safety Population: All participants who received at least 1 dose in Part B.) | 0 | 0 | 53 | 52 | 46 | 45
Completed (All participants who continued from Part A until the End of follow up period.) | 0 | 0 | 55 | 53 | 49 | 49
Not Completed | 0 | 0 | 0 | 0 | 0 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 4
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The analysis was performed on Intent-to Treat (ITT) population which included all randomized participants. Participants were classified according to the treatment as randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Linerixibat 40 Milligrams (mg) | Part A: Placebo | Total
Number analyzed (Participants) | 119 | 119 | 238
Age, Customized [Number; unit: Participants]
  18-49 Years | 42 | 30 | 72
  50-64 Years | 52 | 54 | 106
  >=65 Years | 25 | 35 | 60
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 113 | 226
  Male | 6 | 6 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  HISPANIC OR LATINO | 33 | 21 | 54
  NOT HISPANIC OR LATINO | 85 | 95 | 180
  UNKNOWN | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Part A: Mean Change From Baseline in Monthly Itch Scores Over 24 Weeks Using Numerical Rating Scale (NRS)
Description: Itch Scores were assessed using a NRS twice daily, ranging from 0 to 10, where 0 represents no itching and 10 the worst imaginable itching. The worst daily itch score was defined as the worst of the two scores recorded daily. The weekly itch score was defined as the average of the worst daily itch scores in one week. The monthly itch score was defined as the worst weekly itch score for the month (4 weeks). Higher monthly itch scores indicate worse itching. Baseline is the worst weekly itch score in the 28 days prior to randomization (Day 1). Change from Baseline is defined as the post dose value minus baseline value. Least-squares (LS) means and the corresponding 95% confidence intervals are reported by taking average of LS means of change from baseline in monthly itch scores obtained over 24 weeks using equal weighting for all time points. Analyzed using Mixed Model Repeated Measures (MMRM) method.
Time Frame: Baseline and up to Week 24
Population: The analysis was performed on the Intent to Treat (ITT) set that included all randomized participants. Participants in the ITT Population were classified according to the treatment as randomized.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Part A: Linerixibat 40 Milligrams (mg) | Part A: Placebo
Number analyzed (Participants) | 119 | 118
Scores on a scale | -2.86 [-3.23 to -2.50] | -2.15 [-2.51 to -1.78]
Statistical Analysis 1: Comparison: Part A: Linerixibat 40 Milligrams (mg) vs Part A: Placebo; The mixed model repeated measures analysis includes Treatment Group, Visit, Visit*Treatment Group interaction, Baseline Monthly Itch score (MIS), Visit*Baseline MIS interaction, Baseline Concomitant Itch Medication; Test type: Superiority; p = 0.001, Mixed Models Analysis; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = -0.72, 95% CI 2-sided [-1.15 to -0.28]

2. Secondary Outcome: Part A: Mean Change From Baseline in Weekly Itch Score at Week 2 Using NRS
Description: Itch Score was assessed using a twice daily NRS, ranging from 0 to 10, where 0 represents no itching and 10 the worst imaginable itching. The worst daily itch score was defined as the worst of the two scores recorded daily. The weekly itch score was defined as the average of the worst daily itch scores in one week. Higher weekly itch scores indicate worse itching. Baseline is the average of the Worst Daily Itch scores in the 7 days prior to randomization (Day 1). Change from Baseline is defined as the Week 2 value minus baseline value. Key secondary endpoints were tested in a step-down/hierarchical approach. Mean Change from Baseline in Weekly Itch Score at Week 2 was the first endpoint tested in the hierarchical analysis. LS mean and the corresponding 95% confidence intervals are reported using Mixed Model Repeated Measures (MMRM) method.
Time Frame: Baseline and at Week 2
Population: The analysis was performed on the ITT set that included all randomized participants. Participants in the ITT Population were classified according to the treatment as randomized. Only participants with data at baseline and at least one post-baseline time point were included
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Part A: Linerixibat 40 Milligrams (mg) | Part A: Placebo
Number analyzed (Participants) | 117 | 116
Scores on a scale | -1.78 [-2.08 to -1.48] | -1.07 [-1.37 to -0.77]
Statistical Analysis 1: Comparison: Part A: Linerixibat 40 Milligrams (mg) vs Part A: Placebo; The mixed model repeated measures analysis includes Treatment Group, Week, Week*Treatment Group interaction, Baseline Weekly Itch score (WIS), Visit*Baseline WIS interaction, Baseline Concomitant Itch Medication; Test type: Superiority; p < 0.001, Mixed Models Analysis — Adjusted for multiplicity as per Statistical Analysis Plan (SAP); Mixed Model Repeated Measures Analysis; Mean Difference (Net) = -0.71, 95% CI 2-sided [-1.07 to -0.34]

3. Secondary Outcome: Part A: Mean Change From Baseline in Monthly Sleep Score Over 24 Weeks Using NRS
Description: Sleep Scores were assessed using an NRS scale, ranging from 0 to 10, where 0 represents no sleep interference and 10 is complete sleep interference. The weekly sleep scale is the average of the daily sleep scores for each week. The monthly sleep score was defined as the worst weekly sleep score for the month (4 weeks). Higher monthly sleep scores indicate higher impact on sleep. Baseline is the worst Weekly Sleep Score in the 28 days prior to randomization (Day 1). Change from Baseline is defined as the post dose value minus baseline value. LS means and the corresponding 95% confidence intervals are reported by taking average of LS means of change from baseline in monthly sleep scores obtained over 24 weeks using equal weighting for all time points analyzed using Mixed Model Repeated Measures (MMRM) method. Mean Change from Baseline in Monthly Sleep Score over 24 weeks was the second endpoint tested in the hierarchical analysis.
Time Frame: Baseline up to Week 24
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Part A: Linerixibat 40 Milligrams (mg) | Part A: Placebo
Number analyzed (Participants) | 119 | 118
Scores on a scale | -2.77 [-3.15 to -2.38] | -2.24 [-2.62 to -1.86]
Statistical Analysis 1: Comparison: Part A: Linerixibat 40 Milligrams (mg) vs Part A: Placebo; The mixed model repeated measures analysis includes Treatment Group, Visit, Visit*Treatment Group interaction, Baseline Monthly sleep score (MSS), Visit*Baseline MSS interaction, Baseline Concomitant Itch Medication; Test type: Superiority; p = 0.024, Mixed Models Analysis — Adjusted for multiplicity as per Statistical Analysis Plan (SAP); Mixed Model Repeated Measures Analysis; Mean Difference (Net) = -0.53, 95% CI 2-sided [-0.98 to -0.07]

4. Secondary Outcome: Part A: Percentage of Responders Defined as Achieving More Than or Equal to (>=) 2-point Reduction From Baseline in the Monthly Itch Score at Week 24
Description: Monthly Itch Score was assessed using an NRS, ranging from 0 to 10, where 0 represents no itching and 10 the worst imaginable itching. The Monthly Itch Score was determined from the worst weekly itch score for the month (4 weeks). Baseline is the worst weekly itch score in the 28 days prior to randomization (Day 1). Responders were defined as participants achieving >=2-point reduction (improvement) from baseline in the Monthly Itch Score. Percentage of Responders achieving >= 2-point Reduction from Baseline in the Monthly Itch Score at Week 24 was the third endpoint tested in the hierarchical analysis.
Time Frame: At Week 24
Population: The analysis was performed on the ITT set that included all randomized participants. Participants in the ITT Population were classified according to the treatment as randomized. Percentage values were rounded to the nearest whole number.
Measure: Number; unit: Percentage of participants
Arm/Group | Part A: Linerixibat 40 Milligrams (mg) | Part A: Placebo
Number analyzed (Participants) | 119 | 119
Percentage of participants | 68.0 | 64.0
Statistical Analysis 1: Comparison: Part A: Linerixibat 40 Milligrams (mg) vs Part A: Placebo; Cochran-Mantel-Haenszel (CMH) stratified analysis adjusted for baseline factors: Baseline Itch Severity (Moderate: >=4 and less than [<]7, Severe: >=7); Concomitant cholestatic pruritus treatment regimen (Regimen contains Bile Acid Binding Resin [BABR], Regimen does not contain BABR, No defined treatment). Multiple imputation of missing Monthly itch scores was done before deriving responder definitions. Imputed datasets were analyzed using the CMH method and combined; Test type: Superiority; p = 0.539, Cochran-Mantel-Haenszel — Adjusted for multiplicity as per Statistical Analysis Plan (SAP); Percentage difference = 4.0, 95% CI [-9.0 to 17.0]

5. Secondary Outcome: Part A: Percentage of Responders Achieving >=3-point Reduction From Baseline in the Monthly Itch Score at Week 24
Description: Monthly Itch Score was assessed using an NRS, ranging from 0 to 10, where 0 represents no itching and 10 the worst imaginable itching. The Monthly Itch Score was determined from the worst weekly itch score for the month (4 weeks). Baseline is the worst weekly itch score in the 28 days prior to randomization. Responders were defined as participants achieving >=3-point reduction (improvement) from baseline in the Monthly Itch Score. Percentage of Responders achieving >= 3-point Reduction from Baseline in the Monthly Itch Score at Week 24 was the fourth endpoint to be tested in the hierarchical analysis.
Time Frame: At Week 24
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Part A: Linerixibat 40 Milligrams (mg) | Part A: Placebo
Number analyzed (Participants) | 119 | 119
Percentage of participants | 56.0 | 43.0
Statistical Analysis 1: Comparison: Part A: Linerixibat 40 Milligrams (mg) vs Part A: Placebo; Cochran-Mantel-Haenszel (CMH) stratified analysis adjusted for baseline factors: Baseline Itch Severity (Moderate: >=4 and <7, Severe: >=7); Concomitant cholestatic pruritus treatment regimen (Regimen contains BABR, Regimen does not contain BABR, No defined treatment). Multiple imputation of missing Monthly itch scores was done before deriving responder definitions. Imputed datasets were analyzed using the CMH method and combined; Test type: Superiority; p = 0.043, Cochran-Mantel-Haenszel — Adjusted for multiplicity; two-sided p-values <0.05 were considered to be nominally significant as per SAP; Percentage Difference = 13.0, 95% CI 2-sided [0.0 to 27.0]

6. Secondary Outcome: Part A: Percentage of Responders as Achieving a >=4-point Reduction From Baseline in the Monthly Itch Score at Week 24
Description: Monthly Itch Score was assessed using an NRS, ranging from 0 to 10, where 0 represents no itching and 10 the worst imaginable itching. The Monthly Itch Score was determined from the worst weekly itch score for the month (4 weeks). Baseline is the worst weekly itch score in the 28 days prior to randomization. Responders were defined as participants achieving >=4-point reduction (improvement) from baseline in the Monthly Itch Score. Percentage of Responders achieving >= 4-point Reduction from Baseline in the Monthly Itch Score at Week 24 was the fifth endpoint to be tested in the hierarchical analysis.
Time Frame: At Week 24
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Part A: Linerixibat 40 Milligrams (mg) | Part A: Placebo
Number analyzed (Participants) | 119 | 119
Percentage of participants | 41.0 | 29.0
Statistical Analysis 1: Comparison: Part A: Linerixibat 40 Milligrams (mg) vs Part A: Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.058, Cochran-Mantel-Haenszel — Adjusted for multiplicity; two-sided p-values <0.05 were considered to be nominally significant as per SAP; Percentage Difference = 12.0, 95% CI 2-sided [-0.0 to 24.0]

7. Secondary Outcome: Part A: Mean Change From Baseline in Primary Biliary Cholangitis-40 (PBC-40) Domain Scores at Week 24
Description: PBC-40 is a disease-specific health-related quality of life (HRQoL) questionnaire validated for use in participants with PBC. It consists of 40 questions, which are grouped into 6 domains with 3 to 11 questions per domain. Each question is scored from 1 (least impact) to 5 (greatest impact). For all questions, an answer of "Does/Did not apply" was scored 0. All questions within a domain are summed to obtain individual domain score. Domains were: Symptoms (7 questions) with score range 6 to 35, Itch (3 questions) with score range 0 to 15, Fatigue (11 questions) with score range 11 to 55 , Cognitive (6 questions) with score range 6 to 30 , Emotional (3 questions) with score range 3 to 15 and Social (10 questions) with score range 8 to 50 . Higher scores for individual domains represent poorer quality of life. Baseline is the last assessment prior to the first dose of randomized treatment (Day 1). Change from Baseline was calculated as Week 24 value minus Baseline value.
Time Frame: Baseline up to Week 24
Population: ITT population set included all randomized participants. Participants in the ITT Population were classified according to the treatment as randomized. Number of Participants Analyzed (N) was the maximum number of participants analyzed for any domain, while Number analyzed (n) was the number of participants included in the model for each domain.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Part A: Linerixibat 40 Milligrams (mg) | Part A: Placebo
Number analyzed (Participants) | 95 | 100
Scores on a scale
  Cognitive (score range: 6 to 30): number analyzed (Participants) | 95 | 99
  Cognitive (score range: 6 to 30) | -0.71 [-1.60 to 0.18] | -1.47 [-2.36 to -0.58]
  Emotional (score range: 3 to 15): number analyzed (Participants) | 95 | 99
  Emotional (score range: 3 to 15) | -1.07 [-1.57 to -0.57] | -1.34 [-1.83 to -0.84]
  Fatigue (score range: 11 to 55) | -2.94 [-4.63 to -1.26] | -4.54 [-6.21 to -2.86]
  Itch (score range: 0 to 15) | -3.47 [-4.08 to -2.86] | -2.89 [-3.50 to -2.28]
  Social (score range: 8 to 50): number analyzed (Participants) | 95 | 99
  Social (score range: 8 to 50) | -2.57 [-3.71 to -1.43] | -2.42 [-3.56 to -1.29]
  Symptoms (score range: 6 to 35) | 0.54 [-0.18 to 1.25] | 0.08 [-0.62 to 0.79]
Statistical Analysis 1: Comparison: Part A: Linerixibat 40 Milligrams (mg) vs Part A: Placebo; The mixed model repeated measures analysis includes Treatment Group, Visit, Visit*Treatment Group interaction, Baseline PBC-40 domain scores, Visit*Baseline PBC-40 domain scores interaction, Baseline Concomitant Itch Medication; Test type: Superiority — Cognitive; p = 0.176, Mixed Models Analysis — Not adjusted for multiplicity; two-sided p- values <0.05 were considered to be nominally significant as per SAP; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = 0.76, 95% CI 2-sided [-0.34 to 1.86]
Statistical Analysis 2: Comparison: Part A: Linerixibat 40 Milligrams (mg) vs Part A: Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority — Emotional; p = 0.403, Mixed Models Analysis — Not adjusted for multiplicity; two-sided p- values <0.05 were considered to be nominally significant as per SAP; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = 0.27, 95% CI 2-sided [-0.36 to 0.89]
Statistical Analysis 3: Comparison: Part A: Linerixibat 40 Milligrams (mg) vs Part A: Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority — Fatigue; p = 0.132, Mixed Models Analysis — Not adjusted for multiplicity; two-sided p- values <0.05 were considered to be nominally significant as per SAP; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = 1.59, 95% CI 2-sided [-0.48 to 3.67]
Statistical Analysis 4: Comparison: Part A: Linerixibat 40 Milligrams (mg) vs Part A: Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority — Itch; p = 0.132, Mixed Models Analysis — Not adjusted for multiplicity; two-sided p- values <0.05 were considered to be nominally significant as per SAP; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = -0.58, 95% CI 2-sided [-1.34 to 0.18]
Statistical Analysis 5: Comparison: Part A: Linerixibat 40 Milligrams (mg) vs Part A: Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority — Social; p = 0.836, Mixed Models Analysis — Not adjusted for multiplicity; two-sided p- values <0.05 were considered to be nominally significant as per SAP; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = -0.15, 95% CI 2-sided [-1.57 to 1.27]
Statistical Analysis 6: Comparison: Part A: Linerixibat 40 Milligrams (mg) vs Part A: Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority — Symptoms; p = 0.318, Mixed Models Analysis — Not adjusted for multiplicity; two-sided p- values <0.05 were considered to be nominally significant as per SAP; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = 0.45, 95% CI 2-sided [-0.44 to 1.34]

8. Secondary Outcome: Part A: Mean Change From Baseline in Patient's Global Impression of Severity (PGI-S) Over 24 Weeks
Description: The Patient's Global Impression of Severity (PGI-S) is a patient-reported outcome measure used to assess the severity of symptoms from the participant's perspective. The PGI-S asks participant to rate the severity of their itch in the past 7 days on a single item, using a scale ranging from 0 (absent) to 5 (very severe). Higher score indicates higher severity. Baseline is the last assessment prior to the first dose of randomized treatment for Part A (Day 1). Change from Baseline is defined as the post dose value minus baseline value. LS means and the corresponding 95% confidence intervals are reported by taking average of LS means of change from baseline in PGI-S obtained over 24 weeks using equal weighting for all time points, analyzed using Mixed Model Repeated Measures (MMRM) method.
Time Frame: Baseline and up to Week 24
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Part A: Linerixibat 40 Milligrams (mg) | Part A: Placebo
Number analyzed (Participants) | 114 | 111
Scores on a scale | -1.22 [-1.36 to -1.07] | -0.84 [-0.99 to -0.70]
Statistical Analysis 1: Comparison: Part A: Linerixibat 40 Milligrams (mg) vs Part A: Placebo; The mixed model repeated measures analysis includes Treatment Group, Visit, Visit*Treatment Group interaction, Baseline PGI-S score, Visit*Baseline PGI-S score interaction, Baseline Concomitant Itch Medication; Test type: Superiority; p < 0.001, Mixed Models Analysis — Not adjusted for multiplicity; two-sided p- values <0.05 were considered to be nominally significant as per SAP; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = -0.37, 95% CI 2-sided [-0.55 to -0.20]

9. Secondary Outcome: Part A: Patient's Global Impression of Change (PGI-C) Scores Over 24 Weeks
Description: Patient's Global Impression of Change (PGI-C) was assessed using a 7-level response scale, ranging from 1 (very much improved) to 7 (very much worse). Higher score indicates higher level of change. LS means and the corresponding 95% confidence intervals are reported by taking average of LS means of PGI-C obtained over 24 weeks using equal weighting for all timepoints, analyzed using Mixed Model Repeated Measures (MMRM) method.
Time Frame: Week 4 up to Week 24
Population: The analysis was performed on the ITT set that included all randomized participants. Participants in the ITT Population were classified according to the treatment as randomized. Only participants with data for at least one time point were included.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Part A: Linerixibat 40 Milligrams (mg) | Part A: Placebo
Number analyzed (Participants) | 117 | 116
Scores on a scale | 1.97 [1.74 to 2.20] | 2.46 [2.23 to 2.69]
Statistical Analysis 1: Comparison: Part A: Linerixibat 40 Milligrams (mg) vs Part A: Placebo; The mixed model repeated measures analysis includes Treatment Group, Visit, Visit*Treatment Group interaction, Baseline Concomitant Itch Medication; Test type: Superiority; p < 0.001, Mixed Models Analysis — Not adjusted for multiplicity; two-sided p- values <0.05 were considered to be nominally significant as per SAP; Mixed Model Repeated Measures Analysis; Mean Difference (Net) = -0.49, 95% CI 2-sided [-0.76 to -0.21]

10. Secondary Outcome: Part A: Mean Change From Baseline in Alkaline Phosphatase (ALP) at Week 24
Description: Blood samples were collected at indicated time points for evaluation of ALP. Change from Baseline in ALP at Week 24 was evaluated. Baseline was established using an average of two sets of laboratory values obtained at least 4 weeks apart within 56 days prior to randomization (Day 1). Change from Baseline was calculated as Week 24 value minus Baseline value.
Time Frame: Baseline and Week 24
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: International units per liter (IU/L)
Arm/Group | Part A: Linerixibat 40 Milligrams (mg) | Part A: Placebo
Number analyzed (Participants) | 102 | 107
International units per liter (IU/L) | 10.61 [-8.53 to 29.74] | -8.03 [-26.79 to 10.74]

11. Secondary Outcome: Part A: Mean Change From Baseline in Bilirubin at Week 24
Description: Blood samples were collected at indicated time points for evaluation of Bilirubin. Change from Baseline in total bilirubin at Week 24 was evaluated. Baseline was established using an average of two sets of laboratory values obtained at least 4 weeks apart within 56 days prior to randomization (Day 1). Change from Baseline was calculated as Week 24 value minus Baseline value.
Time Frame: Baseline and Week 24
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Micromoles per Liter (mmol/L)
Arm/Group | Part A: Linerixibat 40 Milligrams (mg) | Part A: Placebo
Number analyzed (Participants) | 102 | 107
Micromoles per Liter (mmol/L) | 1.77 [0.84 to 2.71] | -0.31 [-1.24 to 0.62]

ADVERSE EVENTS:
Time Frame: SAEs were collected from the signing of informed consent until last visit (Week 32) or follow up phone call. AEs were collected from start of treatment until last visit (Week 32) or follow up phone call.
Description: All randomized participants from ITT population (N=238) were included in Part A. One participant in Part A was not included in Safety population (N=237) and 15 participants from ITT Population (N=211) in Part B were not included in Safety population (N=196) as they did not receive study intervention.
Arm/Group | Part A: Placebo | Part A: Linerixibat 40 Milligrams (mg) | Part B: Placebo in Part A and Part B | Part B: Placebo in Part A and Linerixibat 40 mg in Part B | Part B: Linerixibat 40 mg in Part A and Placebo in Part B | Part B: Linerixibat 40 mg in Part A and Part B
All-Cause Mortality (participants affected / at risk) | 0/118 | 0/119 | 0/53 | 0/52 | 0/46 | 0/45
Serious Adverse Events (participants affected / at risk) | 4/118 | 14/119 | 0/53 | 0/52 | 2/46 | 0/45
Other Adverse Events (participants affected / at risk) | 54/118 | 96/119 | 5/53 | 16/52 | 3/46 | 7/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Placebo (N=118) | Part A: Linerixibat 40 Milligrams (mg) (N=119) | Part B: Placebo in Part A and Part B (N=53) | Part B: Placebo in Part A and Linerixibat 40 mg in Part B (N=52) | Part B: Linerixibat 40 mg in Part A and Placebo in Part B (N=46) | Part B: Linerixibat 40 mg in Part A and Part B (N=45)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic disorder (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric mucosal lesion (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Placebo (N=118) | Part A: Linerixibat 40 Milligrams (mg) (N=119) | Part B: Placebo in Part A and Part B (N=53) | Part B: Placebo in Part A and Linerixibat 40 mg in Part B (N=52) | Part B: Linerixibat 40 mg in Part A and Placebo in Part B (N=46) | Part B: Linerixibat 40 mg in Part A and Part B (N=45)
Anaemia (Blood and lymphatic system disorders) | 7 (8) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 6 (6) | 8 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 22 (27) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 5 (6) | 8 (14) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 11 (11) | 9 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 21 (28) | 72 (112) | 3 (3) | 14 (18) | 0 (0) | 6 (12)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 9 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 (9) | 8 (13) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 11 (13) | 12 (17) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 3 (3) | 8 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 4 (4) | 11 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 10 (11) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (9) | 7 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 3 (4) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 4 (5) | 10 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholestatic pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-11-20): https://cdn.clinicaltrials.gov/large-docs/27/NCT04950127/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-08): https://cdn.clinicaltrials.gov/large-docs/27/NCT04950127/SAP_001.pdf